CLINICAL TRIAL: NCT04401475
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of EB05 + SOC Vs. Placebo + SOC in Adult Hospitalized Patients with COVID-19
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Edesa has made the decision to suspend this study solely for business reasons. The study stop is not related to any safety concerns of the product.
Sponsor: Edesa Biotech Inc. (Industry)
Collaborators: JSS Medical Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: EB05-04-2020
Record Dates: First submitted 2020-05-21; First posted 2020-05-26 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: COVID-19; ARDS
Keywords: TLR4; ARDS; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This is a multicenter, randomized, double-blind, placebo-controlled, study to evaluate the safety and efficacy of EB05 in adult hospitalized patients with COVID-19. Following enrollment in the study, eligible subjects will be randomized at a ratio of 1:1 at baseline to receive an infusion of either EB05 or Placebo. In addition to study treatment, all patients will receive SOC treatment per routine care at each participating site. Randomization is stratified by site and baseline WHO COVID-19 severity strata defined as Levels 3-4 and Levels 5-6 for the phase 2 study and Levels 6-7 for the phase 3 study.
  The total follow-up duration of each patient will be until 60-days from treatment with the investigational product. All assessments will take place in-hospital except for the 28-day and 60-day follow-up assessment which will be by telephone if the patient has been discharged before this assessment.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stage 1 (Experimental): Stage 1 (Phase II Study) For 80% power (β = 0.20), at a significance level of 5% (α =0.05) and a 1:1 randomization ratio, a total of 316 (EB05: 158, SOC: 158) evaluable patients will be required. Allowing for 20% attrition a total of 396 patients will be recruited.
  Interventions: Biological: SOC plus 15mg/kg EB05 IV; Other: SOC plus Placebo IV
- Stage 2 (Experimental): Stage 2 (Phase III Study) For a 1:1 ratio of patients treated with EB05 vs. Placebo, a cumulative one-sided alpha of 2.5% and 90% power, to detect an Odds Ratio of 2.00, a total of 586 evaluable patients will be required for Stage 2 (Phase III study). 293 of these will be treated with EB05 + SOC and 293 treated with Placebo + SOC. Allowing for 10% attrition, a total of 644 patients will be enrolled in this Stage.
  Interventions: Biological: SOC plus 15mg/kg EB05 IV; Other: SOC plus Placebo IV

INTERVENTIONS:
Biological: SOC plus 15mg/kg EB05 IV — Standard of care plus single IV infusion of 15mg/kg of EB05.
Other: SOC plus Placebo IV — Standard of care plus a single IV infusion of placebo.

SUMMARY:
COVID-19 patients who develop severe disease often develop acute respiratory distress syndrome (ARDS) as a result of a dysregulated immune response. This in turn stimulates a pro-inflammatory cascade ("cytokine storm") as well as emergency myelopoiesis.

This proinflammatory cascade is activated when viral-mediated cell damage occurs in the lungs, resulting in the release of damage-signaling alarmin molecules such as S100A8/A9 (Calprotectin), HMGB1, Resistin, and oxidized phospholipids. These damage-associated molecular patterns (DAMPs) are recognized by the pattern recognition receptor Toll-Like Receptor 4 (TLR4) found on macrophages, dendritic cells and other innate immune cells and result in additional release of pro-inflammatory molecules. Several recent studies have shown that S100A8/A9 serum levels in hospitalized COVID-19 patients positively correlate with both neutrophil count and disease severity. Taken together the DAMP-TLR4 interaction forms a central axis in the innate immune system and is a key driver of the pathological inflammation observed in COVID-19. We hypothesis that targeting the initial step in the signalling pathways of these DAMPs in innate immunity offers the best hope for controlling the exaggerated host response to SARS-CoV-2 infection.

EB05 has demonstrated safety in two clinical studies (>120 patients) and was able to block LPS-induced (TLR4 agonist) IL-6 release in humans. Given, this extensive body of evidence we believe EB05 could ameliorate ARDS due to COVID-19, significantly reducing ventilation rates and mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥18 years of age at the time of consent.
2. Laboratory-confirmed diagnosis of COVID-19.
3. Hospitalized for COVID-19 related respiratory disease.
4. Patient belongs to one of the following two categories in the nine-point COVID-19 severity scale:

   1. Hospitalized, requiring intubation and mechanical ventilation - Level 6 of the nine-point COVID-19 severity scale.
   2. Hospitalized and intubated with additional organ support - pressors, RRT, ECMO - Level 7 of the nine-point COVID-19 severity scale.
5. For women of childbearing potential involved in any sexual intercourse that could lead to pregnancy: Negative pregnancy test and willingness to use contraceptive (consistent with local regulations) during the study period.
6. Signed informed consent obtained by any patient capable of giving consent, or, when the patient is not capable of giving consent, from his or her legal/authorized representatives.

Exclusion Criteria:

1. The subject is a female who is breastfeeding or pregnant.
2. Known hypersensitivity to EB05 or its excipients.
3. In the opinion of the investigator, death is imminent and inevitable or patient will be discharged within the next 48 - 72 hours, irrespective of the provision of treatment.
4. Experiencing cardiac arrest while hospitalized with COVID-19.
5. Active participation in other immunomodulator or immunosuppressant drug clinical trials.

   a. Participation in COVID-19 antiviral, anticoagulant and convalescent plasma trials may be permitted; however, the decision to enroll a patient who is participating in other clinical trials will be dealt with on a case-by-case basis.
6. Treatment with immunomodulator or immunosuppressant drugs, including but not limited to TNF inhibitors and anti-IL-1 agents within 5 half-lives or 30 days (whichever is longer) before randomization. Except for the following, which are permitted:

   1. Treatment with immunomodulator, or immunosuppressant drugs, such as corticosteroids, as part of SOC for COVID-19
   2. Transplant patients
7. Known other clinical conditions that contraindicate EB05 and cannot be treated or solved according to the judgment of the clinician.
8. Patient has been intubated or mechanically ventilated for more than 72 hours prior to administration of the investigational product.
9. Patient has been intubated and then extubated during the current hospitalization prior to administration of the investigational product.
10. Patient has experienced meaningful clinical improvement in the severity of disease prior to administration of the investigational product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 644 (Estimated)
Dates: Start 2020-11-25 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Mortality rate at Day 28 from IP administration. | 28 days
  For the current study, the primary efficacy outcome measure will be the mortality rate from IP administration. Mortality is the most clinically relevant therapeutic endpoint for this population that is on IMV. The primary endpoint will be assessed at 28-days after treatment initiation.

SECONDARY OUTCOMES:
Proportion of patients with clinical improvement at Day 28 | 28 days
  The proportion of patients with clinical improvement, defined as a decrease of two points or more on the World Health Organization (WHO) 9 - point ordinal scale at Day 28 from IP administration.
  The severity of COVID-19 disease is classified according to the WHO 9-point ordinal scale. The minimum value of 0 is associated with an "uninfected" stage wherein no clinical or virological evidence of infection is present. The maximum value of 8 is associated with death. A higher score reflects a worse outcome.
Proportion of patients with clinical improvement at Day 60 | 60 days
  The proportion of patients with clinical improvement, defined as a decrease of two points or more on the World Health Organization (WHO) 9 - point ordinal scale at Day 60 from IP administration.
  The severity of COVID-19 disease is classified according to the WHO 9-point ordinal scale. The minimum value of 0 is associated with an "uninfected" stage wherein no clinical or virological evidence of infection is present. The maximum value of 8 is associated with death. A higher score reflects a worse outcome.
Mortality rate at Day 60 | 60 days
  The mortality rate at Day 60 from IP administration.

OTHER OUTCOMES:
Number of treatment-emergent adverse events (TEAEs) and serious TEAEs. | 28 and 60 days
  Safety Endpoint: Number of treatment-emergent adverse events (TEAEs) and serious TEAEs.

CONTACTS AND LOCATIONS:
Locations (20):
- United States (7):
  - UCSF Fresno, Fresno, California
  - St. Jude Medical Center/ Providence, Fullerton, California
  - University of Miami Hospital, Coral Gables, Florida
  - Baystate Medical Center, Springfield, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Providence Portland Medical Center, Portland, Oregon
  - West Virginia University Medicine Heart & Vascular Institute, Morgantown, West Virginia
- Canada (13):
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver Coastal Health, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - William Osler Health System, Brampton, Ontario
  - Markham Stouffville Hospital, Markham, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Lakeridge Health, Oshawa, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - CISS Monteregie-Centre, Greenfield Park, Quebec
  - Hôpital Maisonneuve Rosemont, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Hôpital Régional de Rimouski, Rimouski, Quebec

IPD SHARING:
Plan to Share IPD: Undecided